CLINICAL TRIAL: NCT03863483
Title: A Phase II, Prospective, Single-center, Randomized, Controlled Study to Investigate the Efficacy and Safety of Sintilimab or Placebo in Combination With Chemotherapy as Second-line Treatment for Patients With Stage IV Nonsquamous Non-small Cell Lung Cancer With Wild-type EGFR After Failure With Platinum-Containing Chemotherapy
Brief Title: A Study of Sintilimab or Placebo in Combination With Chemotherapy as Second-line Treatment for Patients With Stage IV Nonsquamous Non-small Cell Lung Cancer With Wild-type EGFR After Failure With Platinum-Containing Chemotherapy.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xin-Hua Xu (Other)
Responsible Party: Sponsor-Investigator, Xin-Hua Xu, professor, China Three Gorges University, Yichang, China
Organization: China Three Gorges University, Yichang, China (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTGU003
Record Dates: First submitted 2019-03-04; First posted 2019-03-05 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Nonsquamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — sintilimab; Docetaxel; Pemetrexed

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sintilimab plus chemotherapy (Experimental): Sintilimab (200 mg) plus chemotherapy (physicians' choice between docetaxel and pemetrexed) every 3 weeks.
  Interventions: Drug: Sintilimab; Drug: Docetaxel; Drug: Pemetrexed
- Placebo plus chemotherapy (Active Comparator): Placebo plus chemotherapy (physicians' choice between docetaxel and pemetrexed) every 3 weeks.
  Interventions: Drug: Docetaxel; Drug: Pemetrexed; Drug: Placebo

INTERVENTIONS:
Drug: Sintilimab — Sintilimab will be administered intravenously at a fixed dose of 200 milligrams (mg) on Day 1 of each 21-day cycle.
  Arms: Sintilimab plus chemotherapy
Drug: Docetaxel — Docetaxel 75 milligrams per square meter (mg/m^2) will be administered intravenously on Day 1 of each 21-day cycle.
Drug: Pemetrexed — Pemetrexed 500 mg/m^2 will be administered intravenously on Day 1 of each 21-day cycle.
Drug: Placebo — 0.9% sodium chloride injection as placebo will be administered intravenously at a fixed dose of 100 milliliters (mL) on Day 1 of each 21-day cycle.
  Arms: Placebo plus chemotherapy

SUMMARY:
This prospective, single-center, randomized, controlled study will evaluate the efficacy and safety of sintilimab or placebo in combination with chemotherapy as second-line treatment for patients with stage IV nonsquamous non-small cell lung cancer with wild-type EGFR after failure with platinum-containing chemotherapy. Treatment may continue as long as participants are experiencing clinical benefit as assessed by the investigator, i.e., in the absence of unacceptable toxicity or symptomatic deterioration attributed to disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in clinical research; fully understand and know the research and sign informed consent;
2. Age ≥ 18 years old and ≤ 75 years old, either sex;
3. Eastern Collaborative Oncology Group Performance status (ECOG PS) 0, 1 or 2;
4. Has a histologically or cytologically confirmed diagnosis of stage IV (according to the 8th edition of the International Association for the Study of Lung Cancer) nonsquamous NSCLC;
5. Have at least one measurable lesion as defined by RECIST 1.1;
6. Has progression of disease after treatment with at least two cycles of a platinum-containing doublet chemotherapy according to RECIST V.1.1;
7. Patients without activating EGFR mutation;
8. Normal hepatic function: total bilirubin≤1.5×normal upper limit (ULN); Alanine aminotransferase and Aspartate aminotransferase levels ≤2.5×ULN or ≤5×ULN if liver metastasis is present;
9. Normal renal function: Creatinine ≤1.5×ULN or calculated creatinine clearance ≥45 mL/min (using Cockcroft/Gault formula to calculate );
10. Normal hematological function: absolute neutrophil count ≥1.5×109/L, platelet count ≥70×109/L, hemoglobin≥80g/L [no blood transfusion or erythropoietin (EPO) within 7 days] Dependency];
11. Has a life expectancy of at ≥3 months.

Exclusion Criteria:

1. ECOG PS >2;
2. Small cell lung cancer and squamous NSCLC;
3. EGFR mutation or mutation status unknown;
4. Known hypersensitivity or allergy to monoclonal antibody;
5. Prior therapy with an anti-programmed cell death (PD)-1, anti-PD-L1, anti-PD-L2, anti-tumor necrosis factor CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways);
6. Active autoimmune disease, or a documented history of autoimmune disease;
7. Treatment with systemic corticosteroids (prednisone≥10mg per day or equivalent dose) or other systemic immunosuppressive medications within 2 weeks prior to the first dose;
8. Known history or active human immunodeficiency virus (HIV);
9. Known acute or chronic active hepatitis B (HBV DNA positive) infection or acute or chronic active hepatitis C (HCV antibody positive and HCV RNA positive) infection;
10. Interstitial lung disease, or history of pneumonitis requiring systemic steroids for treatment;
11. Active or poorly controlled severe infection;
12. Have serious cardiovascular disease: Symptomatic congestive heart failure (New York Heart Association grade III-IV), unstable angina pectoris, unstable arrhythmia, myocardial infarction or cerebrovascular accident within 3 months before randomization;
13. Received thoracic radiation therapy of >30 Gy within 6 months prior to first dose of study drug;
14. Completed palliative radiotherapy within 7 days prior to first dose of study drug;
15. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-03-26 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Compare Overall Survival (OS) between sintilimab +chemotherapy and placebo + chemotherapy. | approximately 24 months
  To compare the efficacy of the combination of sintilimab and chemotherapy versus placebo and chemotherapy in terms of overall survival (OS) in patients with stage IV nonsquamous non-small cell lung cancer with wild-type EGFR after failure with platinum-containing chemotherapy. Overall Survival (OS) was defined as the time from the date of randomization to the date of death due to any cause. Data for participants who were not reported as dead at the time of analysis was censored at the date when they were last known to be alive.

SECONDARY OUTCOMES:
Compare objective response rate between sintilimab +chemotherapy and placebo + chemotherapy. | approximately 24 months
  ORR was defined as the percentage of participants with confirmed objective tumor response, complete response (CR) or partial response (PR), as determined by investigator using RECIST v1.1 criteria.
Compare Progression Free Survival (PFS) between sintilimab +chemotherapy and placebo + chemotherapy using RECIST 1.1. | approximately 24 months
  PFS was defined as the time between the date of randomization and the date of first documented disease progression or death, whichever occurs first. Disease progression was determined based on investigator assessment using response evaluation criteria In solid tumors (RECIST) v1.1.
Compare duration of response between sintilimab +chemotherapy and placebo + chemotherapy. | approximately 24 months
  DOR was defined as the duration from the first tumor assessment that supports the participant's objective response (CR or PR, whichever is first recorded) to disease progression or death due to any cause, whichever occurs first.
Number of Participants who Experience Treatment Related Adverse Events (AEs). | approximately 24 months
  All Adverse Events and Serious Adverse events will be collected and collated according to grade and frequency. AEs graded using CTCAE (Version 4.0) criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Central Hospital of Yichang City, the First Clinical Medical College of Three Gorges University, Yichang, Hubei, China

IPD SHARING:
Plan to Share IPD: No